CLINICAL TRIAL: NCT04165382
Title: A Before and After Study for Development, Implementation, and Evaluation of a Clinical Practice Guideline for Care of Preterm Infants Receiving Non-invasive Ventilation (NIV)
Brief Title: Development, Implementation and Evaluation of a Clinical Practice Guideline for Care of Preterm Infants Receiving Non-invasive Ventilation (NIV)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Chan Sin Yee, Nurse Consultant (Neonatal Care), Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KC/KE-19-0093/ER-1
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Noninvasive Ventilation
Keywords: nurse care; non-invasive ventilation; preterm infants
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Usual care will be provided to the study group of the Pre-implementation period, and interventions in the guideline will be started to provide to the study group in the Post-implementation period.
Who Masked: Outcomes Assessor
Masking Description: Masking will be applied to the Assessor who is responsible for auditing nurses' compliances to the guideline in the NICU. The Assessor is asked to perform audits regarding the care to infants receiving NIV in the pre-implementation period and post-implementation period without informing him/her for the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation study group (Other): Preterm infants receiving NIV before the implementation of the guideline
  Interventions: Other: Usual care to infants receiving NIV
- Post-implementation study group (Other): Preterm infants receiving NIV after the implementation of the guideline
  Interventions: Other: Interventions in the guideline to infants receiving NIV

INTERVENTIONS:
Other: Interventions in the guideline to infants receiving NIV — Interventions in the guideline involve six components as
  1. choice of "right" nasal interfaces and bonnet
  2. use of skin protective dressing
  3. alternate the nasal interfaces every 6 hours;
  4. positioning the infants at optimal developmental body position without prone every 4-6 hours, and well supporting the devices to prevent displacement and traction
  5. supportive care with more new interventions
  6. regular assessments on infants receiving NIV for pain level and skin integrity for the areas in contacting with the nasal interfaces and devices of NIV
  Other Names: care bundle of the guideline
  Arms: Post-implementation study group
Other: Usual care to infants receiving NIV — Usual care includes the choice of nasal interface for NIV; use of skin protective dressing; positioning of infants without specific frequency or types of position; supportive care as to provide humidification to the ventilator circuit, to remove water condensate in the ventilator circuit, to provide oral care every 3-4 hours and avoid unnecessary nasal suctioning.
  Other Names: Usual care
  Arms: Pre-implementation study group

SUMMARY:
Non-invasive ventilation (NIV) is increasingly used for supporting preterm infants with respiratory distress in the Neonatal Intensive Care Unit (NICU), and the incidence for nasal injury including skin redness or breakdown associated with pressure from the nasal interfaces is found in infants receiving this support. Risk is found higher in preterm infants than term infants due to the smaller gestation age and lower birth weight. Thus, the study aims to develop, implement, and evaluate an evidence-based practice guideline (the guideline) for preterm infants receiving NIV in the NICU. With the implementation of this guideline, it helps to promote comfort to infants receiving NIV, and at the same time to minimize complications associated with NIV.

DETAILED DESCRIPTION:
A workgroup is formed in the NICU to provide expert opinions in the process of development, implementation, and evaluation of the guideline. It consists of five nurses, one neonatologist and one physiotherapist. After that, 16 evidence-based articles were identified in several scientific databases, and practices in the guideline are developed after reviewed and appraised the articles.

Interventions in the guideline involve six components as

1. choice of "right" nasal interfaces, in which the "right" size of nasal interface either short binasal prongs or nasal mask is chosen according to the size of the infant's nose and distance between two nasal nares. In addition, the "right" size of bonnet using to anchoring the ventilator tubing is also selected according to the size of infant's head.
2. use of skin protective dressing, in which the hydrocolloid dressing is used to cover the skin areas underneath the nasal interface and anchoring straps;
3. alternate the nasal interfaces from the short binasal prongs to nasal mask every 6 hours;
4. positioning the infants regularly for 4-6 hours, at optimal developmental body position but avoid prone position, and well supporting the devices to prevent displacement and traction onto the infant's skin after changed position;
5. supportive care including to wet the prongs with sterile water or saline before inserting into the nasal nares, to clean the infant's faces and nasal areas daily, to wipe away any water condensate over infant's nasal areas every 4-6 hours, to gently massage the areas during removal of the nasal interfaces or devices for examination at every routine care, to provide oral care every 3-4 hours and avoid unnecessary nasal suctioning, to provide adequate humidification to the ventilation circuit, to remove water condensate in the interfaces and ventilator circuit, to aspirate air from the gastric tube before every tube feeding to relieve abdominal distension;
6. regular assessments on infants receiving NIV for pain level by Neonatal Pain, Agitation and Sedation Scale, intact of skin integrity for the areas in contacting with the nasal interfaces and devices of NIV, and to rate the severity of injury by the staging system from National Pressure Ulcer Advisory Panel.

The study includes two periods of "pre-implementation" and "post-implementation". In the pre-implementation period, all infants receiving NIV will be providing the usual care including choice of nasal interfaces in which larger or smaller interfaces may be given to the infant, use of skin protective dressing, positioning which is not restricted to the frequency of turning or types of position, supportive care of providing humidification to the ventilator circuit, oral care and avoiding of unnecessary nasal suctioning, removing of water condensate in the ventilator circuit, aspirating of air before alternate tube feeding.

A one-month training will be given to nurses working in the NICU after completion of the pre-implementation period. The training contains a dialect lecture, video demonstration of care, and scenario discussion.

After completion of the one-month training, the post-implementation period will be commenced, and the care in the guideline will be provided to infants receiving NIV.

Data collection on infant participants and nurses will be conducted during the study period.

Data analysis will be performed to evaluate the effectiveness of the guideline as well as the increase of nurses' knowledge in care of infants receiving NIV and their compliances to the guideline.

ELIGIBILITY:
Inclusion Criteria:

* the infant born before 37 completed weeks of gestation age
* receiving or started NIV via nasal prong or nasal mask at the supports as
* continuous positive airway pressure
* non-invasive intermittent positive pressure ventilation
* neural adjusted ventilatory assisted ventilation

Exclusion Criteria:

* infants with the chromosomal abnormalities (e.g. Pierre Robin Sequence)
* complex heart problems (e.g. transposition of great arteries, Tetralogy of Fallot, Coarctation of Aorta)
* severe respiratory disorders/diseases (e.g. diaphragmatic hernia, tracheoesophageal fistula, cystic fibrosis, congenital cystic adenomatoid malformation)
* craniofacial anomalies (e.g. bilateral cleft lip,cleft palate, choanal atresia)
* congenital skin disorders (e.g. collodion baby)
* severe acute conditions (e.g. necrotizing enterocolitis, pneumothorax, intraventricular haemorrhage, severe sepsis)
* parents or legal guardian refuse to join the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
nasal injury | receiving NIV through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  infant's severity of nasal injury rated by the staging system from National Pressure Ulcer Advisory Panel
pain level | receiving NIV through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  infant's pain level rated by the Neonatal Pain, Agitation and Sedation Scale (N-PASS) with minimum score at 0 and maximum score at 11 for preterm < 30 weeks & 10 for infants > or = 30 weeks. To study whether the interventions of the guideline can promote comfort for preterm infants receiving NIV, by studying indirectly on the pain level. For each infant participant, baseline of pain level will be obtained at the beginning of NIV, then pain score will be assessed every shift or every routine care (at least 4 hours) if the baseline score >3. If the pain score reduce or remain unchanged after implementation of the guideline, it shows the comfort of the infants receiving NIV
activity level | receiving NIV through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  infant's activity level including sleep, active, quiet, irritable and unresponsive evaluated in hourly nursing assessment
body weight | receiving NIV through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  infant's body weight weighed by the baby weight scale every alternate day
abdominal girth | receiving NIV through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  infant's abdominal girth by the measuring tape every morning before feeding

SECONDARY OUTCOMES:
knowledge level of caring infants receiving NIV | once before the training, once just after the training, once at 12-week after completion of the one-month training in the NICU
  self-developed questions as "pre-test" and "post-test" to assess nurses' knowledge of caring infants receiving NIV, the minimum score of the test is 0 and maximum is 10, the differences between the score obtained in "pre-test" and "post-test" indicates any increase of knowledge level of caring infants receiving NIV
Compliance to the guideline | once as baseline record in the pre-implementation period, once at 12-week and once at 24-week since the commencement of post-implementation period
  self-developed audit tool to assess nurses' compliance to the guideline
ventilation day | receiving ventilation support through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  total ventilation days for infant receiving NIV and receiving invasive ventilation before changed to NIV
Efficacy of NIV | receiving NIV through study period completion, an average of 6 months for pre-implementation group, and 8 months for post-implementation group
  study the total ventilation day for infants receiving NIV, and any failure of NIV as indicated by infant requiring intubation for the invasive ventilation within 24-hour after receiving NIV

CONTACTS AND LOCATIONS:
Overall Officials: Sin Yee Chan, Principal Investigator — The Queen Elizabeth Hospital; Janita Chau, Professor, Study Chair — Chinese University of Hong Kong
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No